CLINICAL TRIAL: NCT03181477
Title: Multicenter Phase II Study Evaluating the Efficacy of Radiotherapy With Modulation Intensity and Integrated Boost (SIB-IMRT) at the Dose of 80Gy, Associated With Chemotherapy by Temozolomide in the Treatment of Adult Glioblastomas
Brief Title: Study Evaluating the Efficacy of Radiotherapy With SIB-IMRT, Associated With Temozolomide in Glioblastomas
Acronym: Glio-SIB-Up
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-A000679-42
Record Dates: First submitted 2017-06-07; First posted 2017-06-08 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Glioblastoma, Adult
Keywords: Phase II; Radiotherapy with SIB-IMRT; Tomozolomide
MeSH Terms: conditions — Glioblastoma | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- radiotherapy + chimiotherapy (Other): Radiotherapy of 80 GY + Chemotherapy (Temozolomide)
  Interventions: Device: Radiotherapy

INTERVENTIONS:
Device: Radiotherapy — Radiotherapy of 80 GY + Chemotherapy (Temozolomide)

SUMMARY:
Glioblastoma (GBM) is the most aggressive and most frequent brain tumour. Approximately four people per 100,000 inhabitants are diagnosed with this disease every year. The standard treatment comprises surgical resection (whenever possible), normofractionated radiotherapy at a dose of 60Gray (Gy) and temozolomide (TMZ). Median overall survival in these patients is 14.6 months [13.2-16.8].

In a previous phase I clinical trial, dose escalation tolerance using simultaneous-integrated boost intensity-modulated radiation therapy (SIB-IMRT) technic has been evaluated. The investigator demonstrated that SIB-IMRT until a dose of 80Gy in 32 daily fractions, associated with TMZ is feasible and well tolerated by patients with glioblastoma.

The aim of this present phase II clinical trial is to evaluate the overall survival at 18 months for patients with glioblastoma receiving TMZ, according to standard protocol, associated to radiotherapy delivered at 80Gy using SIB-IMRT technic. The first planning target volume (PTV), including oedema and tumour highlighted on T2 flair magnetic resonance imaging (MRI) sequences, will receive 60.8Gy in 32 daily fractions. The second PTV, including tumour highlighted on T1 MRI sequences, will receive 80.0Gy in 32 daily fractions.

Secondary objectives are tolerance, survival free progression and quality of live evaluations.

Sixty seven patients will be enrolled in this present trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 18 to 70 years old.
* Patients with a unifocal Glioblastoma (grade IV astrocytoma in the World Health Organization (WHO) classification) with postoperative macroscopic residue after biopsy or resection alone.
* Location of the tumor or residual tumor, detected by Magnetic Resonance Imaging (MRI) sequences T1 gadolinium, more than 1cm from the optic chiasm
* Diagnosis confirmed by pathology.
* Time from surgery (if performed) and the start of radiation therapy less than 6 weeks.
* performance status 0 or 1 in the WHO classification.
* methylation status of the MGMT promoter gene requested
* blood count: Neutrophil more than 1500/mm3 Platelets more than 100 000/mm3
* Liver function test Bilirubin less than 1,5 times upper limit transaminases than 3 times upper limit
* patient informed and informed consent signed
* Possibility to trat by radiation withintensity modulated (fixed beams modulated or rotational modulation (TomoTherapy, dynamic arctherapy)) strictly respecting the constraints to organs at risk (Crystalline: 8 Gy max, Posterior chamber of the eye: 45 Gy max , optic nerve: 54 Gy max, chiasm: 54 Gy max, brain Stem: 2% 58 Gy D2 <64 Gy, Dmax <69 Gy spinal cord: 46 Gy max, healthy brain (brain - PTV): 60 Gy max 33%, 50 Gy to 50% and D100 <45 Gy to the brain in toto).
* The patient must be affiliated to a social security scheme.

Exclusion Criteria:

* Other histological "Glioblastoma".
* Excision macroscopically complete individualized on postoperative MRI.
* Patient unable to give consent.
* A patient with against-indication to performed MRI (pacemaker, uncontrollable claustrophobia ...).
* The patient must not have received radiation therapy or previous chemotherapy for this condition.
* Other neoplasia unstabilized and / or treated for less than 5 years.
* Patient already included in another clinical trial with an experimental molecule.
* Inability to submit to medical monitoring testing for geographical, social or psychological.
* Pregnancy or breastfeeding
* Private Person of liberty under supervision or under curatorship
* No affiliation to a social security scheme or medical state aid or the universal medical coverage

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2023-09-02 (Actual); Study Completion 2025-09-02 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 18 months

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - CHU Amiens Picardie, Amiens
  - CHU Besançon, Besançon
  - Centre Georges François Leclerc, Dijon
  - Centre d'oncologie et de radiothérapie, Mâcon
  - Institut de cancérologie de Lorraine, Nancy
  - Paul Strauss, Strasbourg
  - Centre de cancérologie des dentellières, Valenciennes

IPD SHARING:
Plan to Share IPD: No